CLINICAL TRIAL: NCT03534349
Title: Lower Limb Flexibility in Duchenne Muscular Dystrophy: Effects on Functional Performance
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Lütfiye AKKURT, Principal investigator, Hacettepe University
Other Study IDs: GO 16/740
Record Dates: First submitted 2018-05-10; First posted 2018-05-23 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Duchenne Muscular Dystrophy; Performance; Flexibility
Keywords: Duchenne Muscular Dystrophy; lower limb flexibility; performance
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigator investigated the effect of lower limb flexibility on functional performance of children with Duchenne Muscular Dystrophy.

DETAILED DESCRIPTION:
Thirty children whose functional levels were in 1 or 2 according to the Brooke Lower Extremity Functional Classification Scale were included in the study. Flexibilities of hamstrings, hip flexors, tensor fascia latae, and gastrocnemius muscles were evaluated in dominant lower limb. Popliteal angle test, hip flexor flexibility test, tensor fascia latae flexibility test and gastrocnemius flexibility test were used for flexibility asssessments. Functional performance was assessed with 6 Minute Walk Test (6 MWT) and Timed Performance Tests. The correlation between the flexibility of lower limb muscles' and performance tests were examined.

ELIGIBILITY:
Inclusion Criteria:

* Having a Duchenne Muscular Dystrophy diagnosis,
* Being in the ambulatory period and climbing four steps independently,
* To be able to cooperate the physiotherapist's directions,
* Not having any severe contracture in the lower limbs which may prevent assessments,
* Not having any injury or surgery involving the lower limbs during the last 6 months.

Exclusion Criteria:

Children who did not provide these criteria and did not will to participate the study were excluded.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with ambule Duchenne Muscular Dystrophy
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test | 6 Minute
  The 6 Minute Walk Test (6MWT) is a standard test recently used to evaluate functional capacity in neuromuscular diseases, and found to be a safe and valid test that can be performed in Duchenne Muscular Dystrophy

SECONDARY OUTCOMES:
Timed Performance Test | 3 minute
  Timed performance tests such as 10 m walk, Gower's (from supine position to stand up), ascending/descending 4 steps were also performed. During these tests, the child's performance was recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Öznur Tunca Yılmaz, Prof., Study Director — Hacettepe University; İpek Alemdaroğlu Gürbüz, Assoc. Prof., Principal Investigator — Hacettepe University; Ayşe Karaduman, Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)